CLINICAL TRIAL: NCT01450254
Title: Effects of Foot Center of Pressure Manipulation on Hip Biomechanics, Muscle Activation Patterns, and Energy Consumption During Gait in Hip Osteoarthritis Patients
Brief Title: Effects of Foot Center of Pressure Manipulation on Hip Osteoarthritis Patients During Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0091-11-EMC
Record Dates: First submitted 2011-10-03; First posted 2011-10-12 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Hip Osteoarthritis
Keywords: Hip Osteoarthritis; Gait Patterns; Neuromuscular retraining
MeSH Terms: conditions — Osteoarthritis, Hip

ARMS (2):
- Experimental (Experimental): These patients will carry out a therapy program with the study intervention device.
  Interventions: Device: AposTherapy Biomechanical System
- Control (Active Comparator): The patients in this group will not carry out a therapy program with the study intervention device.
  Interventions: Other: Control

INTERVENTIONS:
Device: AposTherapy Biomechanical System — The system is a rehabilitation program implementing a device comprised of four adjustable modular elements attached to foot-worn platforms that are capable of manipulating the foot's center of pressure and applying perturbation training throughout the gait cycle. The device allows for neuromuscular training during dynamic loading.
  Arms: Experimental
Other: Control — No intervention will be prescribed to the control group during participation in the study.
  Arms: Control

SUMMARY:
The purpose of this study is to:

1. Analyze the short-term effects of external center of pressure manipulation of the foot in idiopathic hip osteoarthritis patients during gait on:

   1. Gait parameters (spatiotemporal, kinematic, and kinetic)
   2. Muscle activation patterns of the lower limbs and back
2. Analyze the long-term effects (during the period of one year) of external center of pressure manipulation of the foot in idiopathic hip osteoarthritis patients during gait on:

   1. Gait parameters (spatiotemporal, kinematic, and kinetic)
   2. Motor learning and muscle activation patterns
   3. Energy consumption
   4. Pain, physical function, and quality of life

The hypotheses of the study, in reference to the aforementioned study objectives are:

1. Changes in foot center of pressure will have an immediate effect on gait parameters and muscle activation patterns of the lower limbs and back.
2. Long-term manipulation of foot center of pressure, as a result of a year-long rehabilitation program using the AposTherapy Biomechanical System, will result in improvement in gait parameters, changes in muscle activation patterns as a result of new motor learning, improvement in energy consumption, decrease in pain, improvement in physical function, and improvement in quality of life.

DETAILED DESCRIPTION:
This study is a randomized prospective controlled study assessing the short and long-term effects of external foot center-of-pressure manipulation on gait pattern, muscle activation pattern, energy consumption, physical function, pain, and quality of life. Sixty patients will be recruited for the study and divided randomly into two groups, an experimental group (thirty patients) and a control group (thirty patients). Both groups will be similar with respect to demographic and pathological profiles.

The experimental group will be fitted with a customized biomechanical device worn on the feet (AposTherapy Biomechanical System, AposTherapy - Sports and Medical Technologies Ltd., Hertzlia, Israel). The device is custom calibrated for each patient. The device allows center of pressure manipulation for all phases of the gait cycle and induces controlled perturbation during gait. The immediate effects of the device will be evaluated using center of pressure measurements, three-dimensional gait analysis, and surface electromyography. Following this, patients will be instructed to walk with the device at home on a daily basis according to a customized AposTherapy therapy protocol. They will return to the laboratory for measurements of gait pattern, muscle activation pattern, energy consumption, physical function, pain, and quality of life after three months, six months, and twelve months from the start of the therapy protocol. Data from the analyses will be used to reveal potential changes in the aforementioned measurements as a result of the study intervention.

The control group will carry out the same measurements in the laboratory over the period of one year, however without the biomechanical intervention device.

ELIGIBILITY:
Inclusion Criteria:

* Women age 50 and over with unilateral or bilateral idiopathic hip osteoarthritis

Exclusion Criteria:

* Previous surgery on the lower limbs or back
* Previous musculoskeletal injuries and/or diseases of the lower limbs or back
* Cognitive disabilities and/or inability to cooperate or understand study instructions
* Vestibular problems and/or use of a walking aid
* Neurological and/or orthopaedic and/or cardiovascular and/or pulmonary disorders or risks that may impact the patient's functional performance or limit exercise

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Gait Patterns at 3 months, 6 months, and 12 months | From beginning of patient participation in study, after 3 months, after 6 months, and after 12 months
  Three-dimensional gait analysis of spatiotemporal, kinetic, and kinematic parameters.
  Center of pressure measurements.
Change from Baseline in Muscle Activation Patterns at 3 months, 6 months, and 12 months | From beginning of patient participation in study, after 3 months, after 6 months, and after 12 months
  Surface electromyographic analysis of muscle activation patterns.

SECONDARY OUTCOMES:
Change from Baseline in Physical Function at 3 months, 6 months, and 12 months | From beginning of patient participation in study, after 3 months, after 6 months, and after 12 months
  Self-evaluation questionnaires.
  Physical function tests.
  Energy consumption measurements.
Change from Baseline in Pain at 3 months, 6 months, and 12 months | From beginning of patient participation in study, after 3 months, after 6 months, and after 12 months
  Self-evaluation questionnaires.
Change from Baseline in Quality of Life Assessments at 3 months, 6 months, and 12 months | From beginning of patient participation in study, after 3 months, after 6 months, and after 12 months
  Self-evaluation questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Biorobotics and Biomechanics Lab, Technion Israel Institute of Technology, Haifa, Israel